CLINICAL TRIAL: NCT06570187
Title: The Effect of Dexmedetomidine on the Renal Functions in Septic Critically Ill Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kanzy Mostafa Hassan, Clinical Pharmacist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CL (3635)
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Septic Shock; Acute Kidney Injury
Keywords: Dexmedetomidine; acute kidney injury; sepsis; critically ill patients; sedation; prospective clinical trial
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Intervention Model Description: Participants will be randomly distributed into two groups:
  1. Group one: 64 adult participants receiving standard treatment of sepsis and septic shock with dexmedetomidine.
  2. Group two: 64 adult participants receiving standard treatment of sepsis and septic shock and the standard sedatives without dexmedetomidine.
  Both groups can receive other sedatives as add-ons if needed. Guided by Richmond Agitation and Sedation Scale (RASS) and clinical response.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Participants will receive the standard sepsis and septic shock treatment with dexmedetomidine, which is to be administered with an initial dose of 0.2 μg/kg/hour, and the infusion rate is to be titrated based on response for at least 24 hours.
  Interventions: Drug: Dexmedetomidine
- Control (Active Comparator): Participants will receive the standard sepsis and septic shock treatment and the standard sedatives without dexmedetomidine.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be administered with an initial dose of 0.2 μg/kg/hour, infusion rate is to be titrated based on response for at least 24 hours.
  Arms: Dexmedetomidine
Drug: Propofol — Propofol will be administered as the comparator sedative with the standard treatment of sepsis and septic shock.
  Arms: Control

SUMMARY:
This clinical trial aims to evaluate the effect of dexmedetomidine in Sepsis-Associated Acute Kidney Injury in critically ill patients by answering the following questions:

1. What is dexmedetomidine's effect on kidney functions?
2. What is the safety and efficacy of dexmedetomidine in Sepsis-Associated Acute Kidney Injury?

The investigator will compare dexmedetomidine to the standard sedative.

The Participant will take either dexmedetomidine or the standard sedative during their hospitalization, with follow-up of the following:

1. Vital signs including blood pressure, body temperature, respiratory rate, heart rate, and oxygen saturation.
2. Laboratory data including kidney function tests, electrolytes, complete blood count, and liver function tests.
3. An electrocardiogram will be followed to check the heart's electrical activity.
4. The level of alertness or agitation to avoid over and under-sedation.
5. The level of organ dysfunction and mortality risks.
6. Duration of mechanical ventilation.
7. Duration of hospitalization.

DETAILED DESCRIPTION:
Recently, it has been confirmed that dexmedetomidine has an organ protective effect, including the nervous system, heart, lungs, kidneys, liver, and small intestine. These properties allow dexmedetomidine to be a promising candidate for clinical multiorgan protection.

Aim of the study: Evaluation of the effect of dexmedetomidine in Sepsis-Associated Acute Kidney Injury (SA-AKI).

Objectives:

1. Assessment of dexmedetomidine effect in SA-AKI through following serum creatinine (SCr) level, urinary output (UOP), and the need for renal replacement therapy (RRT).
2. Assessment of dexmedetomidine safety in SA-AKI through following the incidence of new-onset bradycardia, and hypotension requiring intervention.
3. Assessment of dexmedetomidine efficacy by determining the effect on hospital mortality, duration of mechanical ventilation (MV), days free of agitation, incidence of organ dysfunction other than AKI, and length of hospital and ICU stay.

Study Design:

The study will be a prospective, randomized, parallel, controlled, open-label clinical trial including 128 participants with SA-AKI. Participants will be recruited from the Critical Care Department at Cairo University Hospitals. Randomization will be carried out using Random Allocation Software. Patients will be randomly allocated into two groups after screening for inclusion and exclusion criteria.

Written informed consent will be obtained from participants' legal caregivers.

Ethical committee approval will be available.

The primary investigator will be responsible for data collection. Each participant will be presented using a sequential number.

Participants recruitment and concealment allocation, data collection, data management, and data analysis will all be subjected to supervision and on-site auditing by academic and medical supervisors. For data verification, medical records revision will be done, to ensure the accuracy and completeness of the collected data.

Based on the pattern and percentage of missing data, the study investigator is expecting either missing completely at random (MCAR) or missing at random (MAR). Accordingly, multiple imputation (MI) will be implemented to handle missing data.

Normal ranges for lab data will be available.

Study outcomes will be assessed every 48 hours.

Sample size calculation:

Sample size calculation was performed using G power software. The sample size was based on an effect size of 0.5272. A total sample size of 116 patients (58 patients per group) is needed to reject the null hypothesis of equality of means between the control and treatment groups with an 80% power at a 5% significance level (α = 0.05) using two tails t-test.

The effect size was calculated based on the difference in SCr between day 1 and day 3 in septic AKI patients (126.3µmol/L ± 27.6 in day 1 vs. 132.3 µmol/L ± 26.4 in day 3 in the control group vs. 113.2 µmol/L ± 28.9 in day 1 vs. 104.3 µmol/L ± 22.1 in day 3 in the dexmedetomidine group).

Including a dropout ratio of 10%, the final total sample size is 128 patients (64 patients per group).

Statistical analysis:

The collected data will be thoroughly revised, coded, and tabulated, followed by statistical analysis. Qualitative data will be presented as numbers and percentages. Quantitative data will be represented as mean and standard deviation (SD), or median and interquartile range (IQR) according to data distribution. Chi-square test will be used to compare groups regarding non-numerical variables. Independent samples t-test of significance will be used to compare two means.

To compare proportions between two qualitative characteristics, the Chi-square (x2) test of significance will be used.

A P-value of less than 0.05 will be considered statistically significant in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years old
* Patients with sepsis who develop AKI within 48 hours during ICU stay
* Need for sedation due to the need for mechanical ventilation (MV) (both invasive and non- invasive) within 48 hours of AKI

Exclusion Criteria:

* Contraindications to dexmedetomidine including any of the following: severe bradycardia (heart rate (HR) < 50 beats/min), sick sinus syndrome or second-to-third degree atrioventricular block unless a pacemaker is inserted
* Acute myocardial ischemia
* Mean arterial blood pressure < 50 mmHg despite adequate resuscitation and vasopressor therapy at the time of enrollment
* Pregnancy or lactation
* Duration of dexmedetomidine infusion < 24 hours
* Severe valvular heart disease
* Active seizures during this ICU admission requiring benzodiazepines
* Proven or suspected traumatic brain injury, intracranial hemorrhage, stroke, or spinal cord injury

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in serum creatinine (SCr) | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Reduction in SCr ≥ 0.3 mg/dL within ≤ 72 hours. For patients known as acute on top of chronic kidney disease (CKD), decrease in SCr to < 1.5 times the baseline

SECONDARY OUTCOMES:
Incidence of Renal Replacement therapy (RRT) | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Incidence of requiring RRT during hospitalization
Change in Sequential Organ Failure Assessment (SOFA). | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Change in SOFA from baseline
Incidence of agitation | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Number of days free of agitation using Richmond Agitation and Sedation Scale (RASS) (0) to (-2).
Incidence of bradycardia | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Incidence of new onset symptomatic bradycardia (defined as heart rate < 50 beats per minutes requiring intervention e.g. pacing, pharmacological support, or modification of dexmedetomidine).
Incidence of hypotension | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Incidence of hypotension requiring an intervention (fluid administration and/or vasopressor therapy, or dose modification if the patient was already on a vasopressor).
Duration on mechanical ventilation | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Number of days on mechanical ventilation
Length of hospital and ICU stay | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Number of days of hospitalization
Incidence of another organ dysfunction | Assessment will be done at time of randomization then every 48 hours through hospitalization stay, an average of 2 weeks
  Incidence of organ dysfunction other than AKI (defined as: Coagulation, platelet count < 100,000/mm3; Hepatic, total bilirubin > 2 mg/dL; Respiratory, ration between oxygen saturation and fractional inspired oxygen SaO2/FiO2 < 315)
In-hospital mortality | From time of enrolment until date of death, assessed up to 1 month
  Incidence of death

CONTACTS AND LOCATIONS:
Overall Officials: Nirmeen A Sabry, Ph.D, Study Chair — Cairo University; Amany M Mohamed, Ph.D, Study Director — Cairo University; Ramadan M Khalil, MD, Study Director — Cairo University; Kanzy M Hassan, B. Pharm, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Manrique-Caballero CL, Del Rio-Pertuz G, Gomez H. Sepsis-Associated Acute Kidney Injury. Crit Care Clin. 2021 Apr;37(2):279-301. doi: 10.1016/j.ccc.2020.11.010. Epub 2021 Feb 13. PMID 33752856
- [Background] Cobussen M, Verhave JC, Buijs J, Stassen PM. The incidence and outcome of AKI in patients with sepsis in the emergency department applying different definitions of AKI and sepsis. Int Urol Nephrol. 2023 Jan;55(1):183-190. doi: 10.1007/s11255-022-03267-5. Epub 2022 Jul 20. PMID 35859220
- [Background] Zarbock A, Koyner JL, Gomez H, Pickkers P, Forni L; Acute Disease Quality Initiative group. Sepsis-associated acute kidney injury-treatment standard. Nephrol Dial Transplant. 2023 Dec 20;39(1):26-35. doi: 10.1093/ndt/gfad142. PMID 37401137
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Bao N, Tang B. Organ-Protective Effects and the Underlying Mechanism of Dexmedetomidine. Mediators Inflamm. 2020 May 9;2020:6136105. doi: 10.1155/2020/6136105. eCollection 2020. PMID 32454792
- [Background] Heybati K, Zhou F, Ali S, Deng J, Mohananey D, Villablanca P, Ramakrishna H. Outcomes of dexmedetomidine versus propofol sedation in critically ill adults requiring mechanical ventilation: a systematic review and meta-analysis of randomised controlled trials. Br J Anaesth. 2022 Oct;129(4):515-526. doi: 10.1016/j.bja.2022.06.020. Epub 2022 Aug 10. PMID 35961815
- [Background] Hu H, An S, Sha T, Wu F, Jin Y, Li L, Zeng Z, Wu J, Chen Z. Association between dexmedetomidine administration and outcomes in critically ill patients with sepsis-associated acute kidney injury. J Clin Anesth. 2022 Dec;83:110960. doi: 10.1016/j.jclinane.2022.110960. Epub 2022 Oct 19. PMID 36272399
- [Background] Cioccari L, Luethi N, Bailey M, Shehabi Y, Howe B, Messmer AS, Proimos HK, Peck L, Young H, Eastwood GM, Merz TM, Takala J, Jakob SM, Bellomo R; ANZICS Clinical Trials Group and the SPICE III Investigators. The effect of dexmedetomidine on vasopressor requirements in patients with septic shock: a subgroup analysis of the Sedation Practice in Intensive Care Evaluation [SPICE III] Trial. Crit Care. 2020 Jul 16;24(1):441. doi: 10.1186/s13054-020-03115-x. PMID 32678054
- [Background] Duff S, Murray PT. Defining Early Recovery of Acute Kidney Injury. Clin J Am Soc Nephrol. 2020 Sep 7;15(9):1358-1360. doi: 10.2215/CJN.13381019. Epub 2020 Apr 1. No abstract available. PMID 32238366
- [Background] Mehta RL. Renal Recovery After Acute Kidney Injury and Long-term Outcomes: Is Time of the Essence? JAMA Netw Open. 2020 Apr 1;3(4):e202676. doi: 10.1001/jamanetworkopen.2020.2676. No abstract available. PMID 32282043
- [Background] Bai Y, Li Y, Jin J, Cheng M, Zhang S, Yang X, Xu J. Effects of early recovery of renal function on adverse renal outcomes and mortality in patients with acute kidney injury: a systematic review and meta-analysis. Int Urol Nephrol. 2024 Jul;56(7):2421-2430. doi: 10.1007/s11255-024-03974-1. Epub 2024 Mar 7. PMID 38451431
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Hughes CG, Mailloux PT, Devlin JW, Swan JT, Sanders RD, Anzueto A, Jackson JC, Hoskins AS, Pun BT, Orun OM, Raman R, Stollings JL, Kiehl AL, Duprey MS, Bui LN, O'Neal HR Jr, Snyder A, Gropper MA, Guntupalli KK, Stashenko GJ, Patel MB, Brummel NE, Girard TD, Dittus RS, Bernard GR, Ely EW, Pandharipande PP; MENDS2 Study Investigators. Dexmedetomidine or Propofol for Sedation in Mechanically Ventilated Adults with Sepsis. N Engl J Med. 2021 Apr 15;384(15):1424-1436. doi: 10.1056/NEJMoa2024922. Epub 2021 Feb 2. PMID 33528922